CLINICAL TRIAL: NCT00925925
Title: Epigenetic Markers of B-Cell Function in Low Birth Weight Infants
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Christian Con Yost, University of Utah
Other Study IDs: 35580
Record Dates: First submitted 2009-06-18; First posted 2009-06-22 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2012-06

CONDITIONS: Low Birth Weight; Small for Gestational Age; Immunodeficiency
Keywords: Low birth weight; small for gestational age; B-cell function; epigenetics; B1a; B1b; CD19; CD5
MeSH Terms: conditions — Immunologic Deficiency Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be stored as frozen mRNA isolates if parents consent to tissue banking.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal Birth Weight (NBW): Term, healthy infants born at normal birth weights
  Interventions: Other: Cord blood collection for analysis
- Low Birth Weight (LBW): Infants born at > or equal to 34 0/7 weeks with a birth weight at < or equal to 10% for gestational age at birth (Small for Gestational Age, SGA)
  Interventions: Other: Cord blood collection for analysis

INTERVENTIONS:
Other: Cord blood collection for analysis — Cord blood will be collected from the placentas at delivery for analysis

SUMMARY:
Low birth weight (LBW) status (< 10% for gestational age at birth) is associated with increased risk for diseases such as type II diabetes mellitus, hypertension, chronic obstructive pulmonary disease and coronary artery disease in adults, and represents one example of the "fetal onset of adult disease" hypothesis. Recent data strongly associates LBW status with impaired innate and adaptive immunity leading to increased risk for severe infections during adolescence or early adulthood. Animal studies suggest that the ratio of certain B lymphocyte subpopulations, the B1a and B1b cells, determines whether deficits in immunity occur.

This study will determine the ratio of B1b to B1a lymphocyte subpopulations in the cord blood of infants born LBW in the late preterm to term gestations (> 34 weeks at birth) and compare those ratios with those of normal birth weight (NBW) controls in a nested case control study design.

Furthermore, animal studies suggest that the expression patterns of CD5 and CD19 proteins determines the cellular phenotype of the B lymphocyte, that of a B1a or a B1b cell, and that the regulatory regions controlling their expression are epigenetically vulnerable. The investigators will therefore isolate DNA and RNA from both B lymphocyte subpopulations and determine whether epigenetic changes to the regulatory regions of the genes coding for CD5 and CD19 protein expression occur in LBW lymphocyte subpopulations as compared to the lymphocytes from NBW infants.

This proposal will be the first human study to examine epigenetic determination of a maladaptive phenotype following LBW status at birth in a specific cell type leading to a specific impairment of innate and adaptive immunity.

ELIGIBILITY:
Inclusion Criteria:

* Infants delivered at University of Utah Health Sciences Center
* For LBW group:

  * Gestational age > or = to 34 0/7 weeks
  * Birth weight < or = to 10% for gestational age
* For NBW group:

  * Term infant controls delivered without complication
* Adequate cord blood sample obtained directly after birth
* Parents or guardians must have signed informed consent

Exclusion Criteria:

* Infants with major congenital anomalies will be excluded

Max Age: 2 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Term or near-term infants born at less than or equal to 10% normal birth weight for gestation.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2009-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Characterize and compare the Low Birth Weight(LBW) B lymphocyte subtype B1b with that of Normal Birth Weight(NBW) infants. | 2 years

SECONDARY OUTCOMES:
Characterize CD19 and CD5 epigenetic regulation in LBW infants as compared to NBW infants. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Christian C Yost, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States